CLINICAL TRIAL: NCT01816009
Title: Multicentric Study, of Non Inferiority, Randomized, Opened, to Evaluate the Two Durations Effectiveness of Antibiotherapy (6 Weeks Versus 12 Weeks) in the Treatment of Osteo-articular Prostheses Infections, With Prosthetic Change (in 1 Time or 2 Long Times) or Not (Articular Washing)
Brief Title: Treatment of the Infections on Osteo-articular Prostheses by 6 Versus 12 Weeks of Antibiotherapy
Acronym: DATIPO
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Tours (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PHRN09 - LB / DATIPO; 2010-021242-22 (EudraCT Number); A101472-32 (Other: AFSSAPS)
Record Dates: First submitted 2013-03-12; First posted 2013-03-21 (Estimated); Last update posted 2025-12-26 (Actual); Status verified 2017-10

CONDITIONS: Prosthesis-related Infections
Keywords: infection; antibiotic; prosthesis
MeSH Terms: conditions — Prosthesis-Related Infections; Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 6 weeks (Experimental): the duration of antibiotic treatment will be six weeks.
  Interventions: Other: duration of antibiotic treatment
- 12 weeks (Active Comparator): the duration of antibiotic treatment will be 12 weeks.
  Interventions: Other: duration of antibiotic treatment

INTERVENTIONS:
Other: duration of antibiotic treatment — Used antibiotics already have the AMM in this indication

SUMMARY:
The study is a prospective, open randomized, non-inferiority trial with two parallel groups, comparing 6 weeks versus 12 weeks of antibiotic treatment following surgery procedure (debridement and retention, 1-stage or 2 stage exchange).

The duration of the treatment antibiotic of prosthetic joint infections is only based on experts' opinion ; this one varies from 6 weeks to several months according to the customs of the influencer.

The principal aim of this study is to explore the efficacy and safety of 6 weeks versus 12 weeks antibiotic therapy duration, both associated with surgical procedure (debridement and retention of implant, one-stage or two stages exchange), in PJI treatment.

The study concerns 410 men or women of more than 18 years include in 34 centres in France.

The duration of the study is of 4 years.

DETAILED DESCRIPTION:
Although the infection risk following primary hip and knee arthroplasties is less than 2%, prosthetic joint infections (PJI) have become more frequent due to the increasing number of patients undergoing surgery. PJI remains one of the most serious complications of prosthetic joint implantation. Each PJI episode represents substantial morbidity with a 5.3-7.2-fold higher cost than for the initial arthroplasty. The management of PJI almost always necessitates the need for surgical intervention and prolonged courses of intravenous or oral antimicrobial therapy. Despite a significant amount of basic and clinical research in this field, many questions pertaining to the definition of infection as well as diagnosis and management of these infections remain unanswered. The optimal surgical and antibiotic treatment of PJI remains unclear. The infection of implant is difficult to treat. According to the Infectious Diseases Society America recommendations of Osmon et al. in 2012, antibiotic therapy duration varies: 3 months for hip arthroplasties (6 months for total knee arthroplasties) for PJI with arthroplasty retention, and 6 weeks for two-stage exchanges.

Sometimes, excessive antibiotic treatment durations are performed because recommendations are not evidence-based sensu strictu and only based on experts' opinion. Short therapy should be benefit to ecologic and economic impact.

While the usual treatment is by the parenteral route for the first 2-4 weeks, this attitude is not evidence-based either. Up to one-third of patients with PJI may experience antibiotic-related or catheter-related problems during parenteral treatment. The one-stage and two-stage exchange of the infected implant has rather comparable success rate in the surgical management of the PJI (about 90%). Recent no-randomized studies indicate that short antibiotic therapy (6 weeks) seems to be efficient.

Our proposal study is to explore the efficacy and safety of 6 weeks in the treatment of PJI, after a surgical procedure.

The principal aim of this study is to explore the efficacy and safety of 6 weeks versus 12 weeks antibiotic therapy duration, both associated with surgical procedure (debridement and retention of implant, one-stage or two stages exchange), in PJI treatment.

Treatments antibiotics are chosen according to the germ and according to the consensual recommendations. Used antibiotics already have the AMM in this indication.

Eligible patients have at least one symptom relating to the PJI (such pain, sinus tract, inflammatory surgical scar…) and microbiological documentation of PJI.The primary endpoint is the occurrence of clinical cure at month 24. Secondary endpoints are (i) adequate clinical and biological response at months 6 and 12, (ii) incidence of adverse events in the two groups, (iii) oral and/or intravenous antibiotic therapy efficacy.

Randomization is stratified by the anatomical location of the infected joint (hip or knee) and surgical procedure (debridement and retention, 1-stage or 2 stage exchange).

The follow-up consists on periodic clinical examinations, anamnesis and occasionally laboratory or radiological controls.

ELIGIBILITY:
Inclusion Criteria:

* Men or women over 18, presenting at least one of the following clinical signs: pain, fever, dent or flow of scar
* Bacterial infection on osteo-articular prosthesis (hip or knee)
* Documented basterial infection
* Surgical care optimized with prothesis change or articular washing
* Infection requiring an antibiotic treatment by parenteral way Intravenous injection or per bone
* Treatment effective antibiotic begun in the most previously 21 days
* Signed consent

Exclusion Criteria:

* Patient with no proof of osteo-articular infection
* No surgical care
* Patient having more than one prothesis change because of sepsis
* Infection due to mycobactery, fungic infection or brucellienne infection
* Patient with life expectancy supposed lower than 2 years
* Guardianship patient
* Patient included in another study

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 410 (Actual)
Dates: Start 2011-11 (Actual); Primary Completion 2017-01-21 (Actual); Study Completion 2017-01-21 (Actual)

PRIMARY OUTCOMES:
occurrence of clinical cure | two years
  Percentage of success in 2 years defined by the absence of infection or relapse in the same germ, and the absence of clinical, biological and radiological signs some of infection (pain, fever). This criterion will be estimated beyond the first 6 weeks of treatment antibiotic after the introduction of the treatment and until 2 years after the stop of the treatment.

SECONDARY OUTCOMES:
microbiological success | 2 years
  negativity of the microbiological samples during second step of 2 stage exchange (in the case of two-stage exchange of the implant).

CONTACTS AND LOCATIONS:
Locations (37):
- France (37):
  - Service de chirurgie orthopédique et traumatologique, CHU d'AMIENS, Amiens
  - Service des maladies infectieuses et tropicales, CHU d'ANGERS, Angers
  - Département de Médecine Interne et Maladies Infectieuses, hôpital privé d'Antony, Antony
  - Service des maladies infectieuses et tropicales, CHU de BESANCON, Besançon
  - Service de médecine interne, CH de BEZIERS, Béziers
  - Service de chirurgie orthopédique et traumatologique, Polyclinique de BLOIS, Blois
  - Service de Maladies Infectieuses et de Médecine Tropicale, Hôpital Pellegrin, CHU de Bordeaux, Bordeaux
  - Service de chirurgie orthopédique et traumatologique, CH de BOURG EN BRESSE, Bourg-en-Bresse
  - Service de Maladies Infectieuses, CH de BOURG EN BRESSE, Bourg-en-Bresse
  - Service de médecine interne et de maladies infectieuses, CHU de BREST, Brest
  - Service des maladies infectieuses et tropicales, CHU de CAEN, Caen
  - Service des maladies infectieuses et tropicales - médecine interne, CH de CHAMBERY, Chambéry
  - Service de médecine interne, rhumatologie, Centre Hospitalier Chalon sur Saône William Morey, Châlon Sur Saone
  - Service de Chirurgie Orthopédique et Traumatologique, APHP Hôpital Antoine Béclère, Clamart
  - Service de Médecine Interne et Immunologie Clinique, APHP Hôpital Antoine Béclère, Clamart
  - Service des maladies infectieuses et tropicales, CH de CLERMONT-FERRAND, Clermont-Ferrand
  - Centre de chirurgie orthopédique et de la main, CHRU de STRASBOURG, Illkirch-Graffenstaden
  - Unité de Traumatologie -Orthopédie septique, CHRU de LILLE, Lille
  - Service de Maladies Infectieuses, CHU de LIMOGES, Limoges
  - Centre de vaccinations internationales et de médecine des voyages du Tonkin, Lyon
  - Service des Maladies Infectieuses et tropicales, CHU de MONTPELLIER, Montpellier
  - Service des Maladies Infectieuses et tropicales, CHU de NANCY, Nancy
  - Service des maladies infectieuses et tropicales Hôtel-Dieu, CHU de Nantes, Nantes
  - Service de Chirurgie orthopédique Hôpital Lariboisière, Paris
  - Service des maladies infectieuses et tropicales CH Saint-Jean, Perpignan
  - Service de médecine interne, maladies infections et tropicales, CHU de POITIERS, Poitiers
  - Service de médecine interne, PONTOISE, Pontoise
  - Service des maldies infectieuses, CH d'ANNECY, Pringy
  - Service de Maladies Infectieuses, CHU de REIMS, Reims
  - Service des Maladies Infectieuses, CHU de RENNES, Rennes
  - Service de pneumologie - maladies infectieuses et tropicales, CH de ST QUENTIN, Saint-Quentin
  - Service d'infectiologie, CH de TOULON, Toulon
  - Service de Chirurgie Orthopédique et Traumatologique, Toulouse
  - Service des maladies infectieuses CH Gustave Dron, Tourcoing
  - Service de Chirurgie Orthopédique et traumatologie, hôpital Trousseau, Tours
  - Service de Médecine Interne et de Maladies Infectieuses, CHRU de TOURS, Tours
  - Service de chirurgie orthopédique, CH de VERSAILLES, Versailles

REFERENCES:
- [Result] Bernard L, Arvieux C, Brunschweiler B, Touchais S, Ansart S, Bru JP, Oziol E, Boeri C, Gras G, Druon J, Rosset P, Senneville E, Bentayeb H, Bouhour D, Le Moal G, Michon J, Aumaitre H, Forestier E, Laffosse JM, Begue T, Chirouze C, Dauchy FA, Devaud E, Martha B, Burgot D, Boutoille D, Stindel E, Dinh A, Bemer P, Giraudeau B, Issartel B, Caille A. Antibiotic Therapy for 6 or 12 Weeks for Prosthetic Joint Infection. N Engl J Med. 2021 May 27;384(21):1991-2001. doi: 10.1056/NEJMoa2020198. PMID 34042388